CLINICAL TRIAL: NCT01257100
Title: Environmental and Genetic Determinants of NPC
Status: Terminated | Type: Observational
Why Stopped: Determined not to be Human Subject Research
Sponsor: National Cancer Institute (NCI) (NIH)
Collaborators: Academia Sinica, Taiwan (Other); National Taiwan University Hospital (Other); Koo Foundation Sun Yat-Sen Cancer Center (Other); Mackay Memorial Hospital (Other); Far Easter Memorial Hospital (Unknown); Cathay General Hospital (Other)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999911040; 11-C-N040
Record Dates: First submitted 2010-12-08; First posted 2010-12-09 (Estimated); Last update posted 2020-06-04 (Actual); Status verified 2020-06

CONDITIONS: Nasopharyngeal Neoplasms; Herpesvirus 4, Human
Keywords: Nasopharyngeal Carcinoma; Epstein-Barr Virus; NPC
MeSH Terms: conditions — Nasopharyngeal Neoplasms; Epstein-Barr Virus Infections; Nasopharyngeal Carcinoma

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other

GROUPS / COHORTS (2):
- Cases with NPC: Cases with NPC
- Hospital based controls: Hospital based controls

SUMMARY:
Background:

- Nasopharyngeal carcinoma (NPC) a common malignant tumor in southern China and Southeast Asia. Infection with Epstein-Barr virus is believed to be necessary for the development of NPC; non-viral environmental factors, such as dietary consumption of nitrosamines, cigarette smoking, betel nut chewing, wood dust exposure and possibly exposure to formaldehyde, have been implicated in the disease. Genetic susceptibility may also play an important role in the development of NPC. However, more information is needed on the connections between genetic and environmental factors in NPC, particularly in areas where the cancer risk appears to be greatest.

Objectives:

- To examine the main effects of genetic factors and environmental exposures (e.g., cigarette smoking, betel nut chewing, formaldehyde, wood dust) on nasopharyngeal carcinoma risk.

Eligibility:

* Cases: Individuals at least 21 years of age who have been diagnosed with NPC at one of the participating hospitals and have been residents of northern Taiwan for at least 6 months.
* Controls: Hospital patients with diseases other than NPC at least 21 years of age, matched to NPC patients based on hospital, age at diagnosis, gender, and ethnicity.

Design:

* This study involves a risk factor interview, medical record abstraction and biological sample collection.
* Participants will respond to interview questions about their lifestyle and risk factors thought to be involved in NPC development.
* All participants will provide blood and saliva samples for study. Participants who have been diagnosed with NPC will also provide consent to allow researchers to study tissue samples taken during tumor biopsies or surgeries.
* Treatment will not be provided as part of this protocol.

DETAILED DESCRIPTION:
Nasopharyngeal carcinoma (NPC) is one of the most common malignant tumors in southern China and Southeast Asia. While infection with Epstein-Barr Virus (EBV) is believed to be necessary for the development of NPC, non-viral environmental factors have also been implicated in the carcinogenesis of NPC including consumption of salted fish and other nitrosamine containing preserved foods, formaldehyde and wood dust exposure, cigarette smoking, and betel nut chewing. In addition to environmental factors, it is widely accepted that genetic susceptibility plays an important role in the pathogenesis of NPC. Polymorphisms in genes involved in antigen presentation, nitrosamine metabolism and DNA repair have been suggested to be associated with NPC risk, and various chromosomal regions linked to NPC development have been reported. Two recently completed NPC GWAS have reported that the strongest evidence for disease association is observed for SNPs located on the 3.6 Mb Major Histocompatibility Complex (MHC) region on chromosome 6p21 where human leukocyte antigen (HLA) genes are located. These associations highlight the role of both environmental exposures and genomic variation in the etiology of NPC. However, the specific role of EBV on NPC pathogenesis is not completely understood and studies to date have had difficulty pinpointing the specific genetic factors involved in NPC pathogenesis due to the complexity of the MHC region and limited sample size of candidate gene studies.

DCEG investigators and their Taiwan colleagues have a longstanding history of studies to elucidate the role of environmental and genetic factors associated with NPC. A case-control study (375 cases; 327 controls) was conducted in the early 1990s and was followed by a large multiplex family study that was completed in 2006 (358 families; 3,216 individuals). Results from these studies have provided a substantial portion of the epidemiological evidence regarding factors linked to NPC development to date.

At this time, we propose a new case-control study in Taiwan designed to 1) comprehensively evaluate environmental risk factors for NPC; 2) systematically evaluate genetic risk factors for NPC for which previous GWAS and candidate-gene studies have suggested an association; and 3) explore gene-gene and gene-environment interactions for strong main effects identified in our study. In total, up to 2000 cases and 2000 controls are expected to be recruited from five participating hospitals in Northern Taiwan. Cases will consist of 550 incident cases ascertained retrospectively and 1350 incident cases ascertained prospectively. Controls will be hospital based; they will be frequency matched (1:1) to cases on age, gender and ethnicity, and will exclude individuals referred to the participating hospitals due to conditions associated with known NPC risk factors.

This project is a collaborative effort between investigators in Taiwan and at the NCI. Investigators in Taiwan will fund the field recruitment and data collection effort. Results from this study have the potential to further clarify currently controversial environmental risk factors as well as elucidate genetic factors of NPC.

ELIGIBILITY:
* INCLUSION CRITERIA:

Eligibility criteria for cases:

* Incident diagnosis of NPC between 2010-2015
* Age greater than or equal to 21 years at NPC diagnosis
* Histologically confirmed
* Resident of northern Taiwan greater than or equal to 6 months

Eligibility criteria for controls:

* Resident of northern Taiwan greater than or equal to 6 months
* Matched to case based on age at diagnosis, gender, and ethnicity

EXCLUSION CRITERIA:

Exclusion criteria for controls:

- Clinic attendance due to conditions associated with EBV or smoking

Ages: 21 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This is a hospital based case control population
Sampling Method: Non-Probability Sample
Enrollment: 3500 (Actual)
Dates: Start 2010-12-08 (Actual); Primary Completion 2020-06-02 (Actual); Study Completion 2020-06-02 (Actual)

PRIMARY OUTCOMES:
Nasopharyngeal carcinoma
  NPC diagnosis

CONTACTS AND LOCATIONS:
Overall Officials: Allan Hildesheim, Ph.D., Principal Investigator — National Cancer Institute (NCI)
Locations (6):
- Taiwan (6):
  - Academia Sinica 128 Academia Road, Taipei
  - Cathay General Hospital 280 Renai Rd, Section 4, Taipei
  - Far Easter Memorial Hospital 21, NanYa S. Rd, Section 2, Ban-Chiao, Taipei
  - Koo Foundation Sun Yat-Sen Cancer Center, Taipei
  - MacKay Memorial Hospital No 92, Section 2, Zhongshan N. Rd, Zhongshan Dist, Taipei
  - National Taiwan University Hospital, Taipei

REFERENCES:
- [Background] Armstrong RW, Imrey PB, Lye MS, Armstrong MJ, Yu MC, Sani S. Nasopharyngeal carcinoma in Malaysian Chinese: salted fish and other dietary exposures. Int J Cancer. 1998 Jul 17;77(2):228-35. doi: 10.1002/(sici)1097-0215(19980717)77:23.0.co;2-7. PMID 9650558
- [Background] Bei JX, Li Y, Jia WH, Feng BJ, Zhou G, Chen LZ, Feng QS, Low HQ, Zhang H, He F, Tai ES, Kang T, Liu ET, Liu J, Zeng YX. A genome-wide association study of nasopharyngeal carcinoma identifies three new susceptibility loci. Nat Genet. 2010 Jul;42(7):599-603. doi: 10.1038/ng.601. Epub 2010 May 30. PMID 20512145
- [Background] Blair A, Saracci R, Stewart PA, Hayes RB, Shy C. Epidemiologic evidence on the relationship between formaldehyde exposure and cancer. Scand J Work Environ Health. 1990 Dec;16(6):381-93. doi: 10.5271/sjweh.1767. PMID 2284588